CLINICAL TRIAL: NCT04296357
Title: Follow-up of Children Born From In-vitro Maturation Versus In-vitro Fertilization: Follow-up of a Randomized Controlled Trial
Brief Title: Health of IVF Versus IVM Children (FM-BABIES)
Acronym: FM-BABIES
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CS/BVMĐ/20/05
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Infertility; IVF; IVM
Keywords: IVF; IVM; ASQ-3; Health of children
MeSH Terms: conditions — Infertility | interventions — Health Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVF children: Children born from in-vitro fertilization
  Interventions: Diagnostic Test: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Diagnostic Test: Developmental Red flags
- IVM children: Children born from in-vitro maturation
  Interventions: Diagnostic Test: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Diagnostic Test: Developmental Red flags

INTERVENTIONS:
Diagnostic Test: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 — Ages & Stages Questionnaires®, Third Edition (ASQ®-3) is a developmental screening tool designed for use by early educators and health care professionals. It relies on parents as experts, is easy-to-use, family-friendly and creates the snapshot needed to catch delays and celebrate milestones.
Other: Physical development and General Health — Physical development and General health examination
Diagnostic Test: Developmental Red flags — Developmental Red flags Questionnaires

SUMMARY:
The investigators conduct a follow up of our randomized controlled trial (RCT) to investigate the development of children born from In-vitro fertilization (IVF) and In-vitro maturation (IVM), in order to give strong evidence about the safety of IVM in women with high antral follicle count or especially polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Since the birth of the first baby born from in-vitro maturation (IVM) in 1991, this technique has been considered an alternative solution for treating infertility beside conventional controlled ovarian stimulation for in-vitro fertilization (IVF). Since then, there are already more than 5000 children born from IVM, and that number is on the trend of increasing.

Regarding technique, immature oocytes (germinal vesicle - GV) were aspirated from secondary follicles sized from 2-10mm, under follicle-stimulating hormone (FSH) priming or no ovarian stimulation at all. Afterward, the maturation process was undertaken in an artificial medium, out of a living body. This technique, by reducing the usage of external hormones, is highly effective in minimizing the risk of ovarian hyperstimulation syndrome (OHSS) in women with high antral follicle count, especially polycystic ovarian syndrome, with a rate of OHSS recorded as low as 0 percent. Alongside that, the pregnancy rate, as well as the live birth rate of IVM, when proceeded well, is not lower than conventional IVF. Until now, there is only one randomized controlled trial comparing these two techniques directly.

Due to differences in the process of culturing between IVM and IVF, primarily the maturation is undertaken in an artificial medium, the health of children born from IVM received many interests. Numerous studies have been conducted to compare the development of children born from IVM and IVF. Neonatal outcomes of children born from IVM and IVF are considerably comparable. And the development of children born from these two techniques is not significantly different. All the information, as mentioned above, was not from randomized controlled trials but retrospective or prospective cohort studies. Thus, we conduct a follow up of our RCT to investigate the development of children born from IVM and IVM, to give strong evidence about the safety of IVM in women with high antral follicle count or especially PCOS.

ELIGIBILITY:
Inclusion Criteria:

* All live babies born following the In-vitro Maturation and In-vitro fertilization from our FM study.
* Parents agree to participate in the study.

Exclusion Criteria:

* Babies died under or at 24 months

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Live babies born following the IVF and IVM from our FM study (NCT03405701)
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
The average total ASQ-3 score | Up to 24 months after birth
  ASQ-3 (Ages and Stages Questionaires®) has 5 aspects: Communication, Gross motor, Fine motor, Problem solving and Personal-Social Each aspect has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  ASQ-3 average = average score of 5 aspects.

SECONDARY OUTCOMES:
Score of Communication | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Gross motor | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Fine motor | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Problem solving | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Personal-Social | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
The rate of children who have at least one red flag sign | From 6 months to 24 months after birth
  He or she has at least one red flag sign by age For children at 6 months: he or she
  * Do not know to flip before 3 months
  * Still holding hands constantly at 3 months
  * Do not pay attention to the stimulation from the environment
  * Poor head control
  * No access to objects/ toys before 5 months
  * No laughter
  For children at 12 months: he or she
  * No babbling before 6 months
  * Unable to sit down in a W-style at 7 months
  * Unable to identify audio source before 10 months
  * Still holding things in your mouth often for 12 months
  For children at 24 months: he or she
  * Do not speak consonants before 15 months
  * Do not know imitate before 16 months
  * Do not know to point fingers to attract attention about objects that he or she cares about
  * Show right-handedness before 18 months
  * Unable to ascend and descend stairs at 24 months
  * Repeat the machinery of others' words
  * Not reached the single 50 marks yet by 24 months
Duration of breast-feeding | Up to 24 months after birth
  Duration of breast-feeding
Infant age at which weaning starts | Up to 24 months after birth
  Infant age at which weaning starts
Name of diseases that lead to hospital admission | Up to 24 months after birth
  Name of diseases that lead to hospital admission
Number of hospital admission | Up to 24 months after birth
  Number of hospital admission
Weight | Up to 24 months after birth
  Weight on the examination date
Height | Up to 24 months after birth
  Height on the examination date

OTHER OUTCOMES:
Gestational age at delivery | At birth
  Gestational age at delivery
Mode of delivery | At birth
  Vaginal birth or C-section
Birth weight | At birth
  Weight of baby born
Length circumference | At birth
  Head circumference after birth Head circumference after birth Head circumference after birth Length circumference after birth
Head circumference | At birth
  Head circumference after birth
Rate of congenital anomalies | At birth
  Any congenital anomalies detected in baby born
Length of neonatal intensive care unit (NICU) admission | Up to 28 days after birth
  Number of admission days to NICU
Rate of Respiratory distress syndrome | Up to 28 days after birth
  Respiratory distress syndrome (RDS), diagnosed as the presence of tachypnoea >60/minute, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram
Rate of Periventricular haemorrhage | Up to 28 days after birth
  Periventricular haemorrhage II B or worse, will be diagnosed by repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al.
Rate of Necrotizing enterocolitis | Up to 28 days after birth
  Necrotizing enterocolitis (NEC) will be diagnosed according to Bell.
Rate of Proven sepsis | Up to 28 days after birth
  Proven sepsis, will be diagnosed on the combination of clinical signs and positive blood cultures.
Rate of Composite of poor perinatal outcomes | Up to 28 days after birth
  Composite of poor perinatal outcomes, defined as intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis or neonatal sepsis.
The rate of long-term illness and chronic conditions | Up to 24 months after birth
  Any long-term illness and chronic condition appears in a child

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vuong LN, Ho VNA, Ho TM, Dang VQ, Phung TH, Giang NH, Le AH, Pham TD, Wang R, Norman RJ, Smitz J, Gilchrist RB, Mol BW. Effectiveness and safety of in vitro maturation of oocytes versus in vitro fertilisation in women with high antral follicle count: study protocol for a randomised controlled trial. BMJ Open. 2018 Dec 9;8(12):e023413. doi: 10.1136/bmjopen-2018-023413. PMID 30530584
- [Result] Cha KY, Koo JJ, Ko JJ, Choi DH, Han SY, Yoon TK. Pregnancy after in vitro fertilization of human follicular oocytes collected from nonstimulated cycles, their culture in vitro and their transfer in a donor oocyte program. Fertil Steril. 1991 Jan;55(1):109-13. doi: 10.1016/s0015-0282(16)54068-0. PMID 1986950
- [Result] Das M, Son WY, Buckett W, Tulandi T, Holzer H. In-vitro maturation versus IVF with GnRH antagonist for women with polycystic ovary syndrome: treatment outcome and rates of ovarian hyperstimulation syndrome. Reprod Biomed Online. 2014 Nov;29(5):545-51. doi: 10.1016/j.rbmo.2014.07.019. Epub 2014 Aug 12. PMID 25262236
- [Result] Gremeau AS, Andreadis N, Fatum M, Craig J, Turner K, McVeigh E, Child T. In vitro maturation or in vitro fertilization for women with polycystic ovaries? A case-control study of 194 treatment cycles. Fertil Steril. 2012 Aug;98(2):355-60. doi: 10.1016/j.fertnstert.2012.04.046. Epub 2012 May 31. PMID 22658347
- [Result] Ho VNA, Braam SC, Pham TD, Mol BW, Vuong LN. The effectiveness and safety of in vitro maturation of oocytes versus in vitro fertilization in women with a high antral follicle count. Hum Reprod. 2019 Jun 4;34(6):1055-1064. doi: 10.1093/humrep/dez060. PMID 31111879
- [Result] Mostinckx L, Segers I, Belva F, Buyl R, Santos-Ribeiro S, Blockeel C, Smitz J, Anckaert E, Tournaye H, De Vos M. Obstetric and neonatal outcome of ART in patients with polycystic ovary syndrome: IVM of oocytes versus controlled ovarian stimulation. Hum Reprod. 2019 Aug 1;34(8):1595-1607. doi: 10.1093/humrep/dez086. PMID 31347678
- [Result] Roesner S, von Wolff M, Elsaesser M, Roesner K, Reuner G, Pietz J, Bruckner T, Strowitzki T. Two-year development of children conceived by IVM: a prospective controlled single-blinded study. Hum Reprod. 2017 Jun 1;32(6):1341-1350. doi: 10.1093/humrep/dex068. PMID 28387798
- [Result] Sauerbrun-Cutler MT, Vega M, Keltz M, McGovern PG. In vitro maturation and its role in clinical assisted reproductive technology. Obstet Gynecol Surv. 2015 Jan;70(1):45-57. doi: 10.1097/OGX.0000000000000150. PMID 25616347
- [Result] Shu-Chi M, Jiann-Loung H, Yu-Hung L, Tseng-Chen S, Ming-I L, Tsu-Fuh Y. Growth and development of children conceived by in-vitro maturation of human oocytes. Early Hum Dev. 2006 Oct;82(10):677-82. doi: 10.1016/j.earlhumdev.2006.01.012. Epub 2006 May 11. PMID 16690233
- [Result] Yu EJ, Yoon TK, Lee WS, Park EA, Heo JY, Ko YK, Kim J. Obstetrical, neonatal, and long-term outcomes of children conceived from in vitro matured oocytes. Fertil Steril. 2019 Oct;112(4):691-699. doi: 10.1016/j.fertnstert.2019.05.034. Epub 2019 Jul 29. PMID 31371040
- [Derived] Vuong LN, Nguyen MHN, Nguyen NA, Ly TT, Tran VTT, Nguyen NT, Hoang HLT, Le XTH, Pham TD, Smitz JEJ, Mol BW, Norman RJ, Ho TM. Development of children born from IVM versus IVF: 2-year follow-up of a randomized controlled trial. Hum Reprod. 2022 Jul 30;37(8):1871-1879. doi: 10.1093/humrep/deac115. PMID 35595193